CLINICAL TRIAL: NCT03894813
Title: Department of Obstetrics and Gynecology, Peking University Shenzhen Hospital
Brief Title: Probiotics as Adjuvant Treatment for Bacterial Vaginosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Collaborators: BGI, China (Other)
Responsible Party: Principal Investigator, Shangrong Fan, Departmemt of Obstetrics and Gynecology, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUshenzhenH2018-016
Record Dates: First submitted 2019-03-14; First posted 2019-03-29 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Probiotics; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics and Metronidazole (Experimental): Probiotics: Oral probiotics(Umeta-Miyue, Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14) ) (qd, 30 days); Metronidazole: Metronidazole vaginal suppositories (qd,7 days)
  Interventions: Drug: "Probiotics" and "Metronidazole"
- Metronidazole vaginal (Active Comparator): Metronidazole vaginal suppositories(1 suppositories,qd,7 days )
  Interventions: Drug: Metronidazole Vaginal

INTERVENTIONS:
Drug: "Probiotics" and "Metronidazole" — Oral probiotics (Umeta-Miyue, Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14) (qd, 30 days)+Metronidazole Suppositories (qd, 7 days)
  Other Names: Umeta-Miyue, Lactobacillus rhamnosus GR-1 & Lactobacillus reuteri RC-14 and Metronidazole Suppositories
  Arms: Probiotics and Metronidazole
Drug: Metronidazole Vaginal — Metronidazole Suppositories,qd, 7 days
  Other Names: Metronidazole Suppositories
  Arms: Metronidazole vaginal

SUMMARY:
The investigators are trying to determine if oral probiotics (Umeta-Miyue, Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14) (30 days)with metronidazole vaginal suppositories(7 days) is better than using metronidazole vaginal suppositories only in preventing the recurrence of bacterial vaginosis (BV).

DETAILED DESCRIPTION:
Studies have shown that oral probiotics can significantly promote the recovery of vaginal flora mainly because intestinal microbiota can migrate and affect vaginal microecology. This project aims to evaluate the efficacy of oral probiotics (Umeta-Miyue, Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14) (30 days) with metronidazole vaginal suppositories(7 days) in the treatment of bacterial vaginosis and to explore the correlation between vaginal flora and fecal flora by detecting the metagenomics of vaginal secretions and intestinal feces at the time of baseline phase, the first month after treatment, the third month after treatment and the sixth month after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years old, with history of sexual activity, premenopausal women；
2. Nugent Score ≥ 7 for diagnosing BV；
3. Sign informed consent.

Exclusion Criteria:

1. mixed vaginitis, such as vulvovaginal candidiasis (VVC), Trichomonas vaginalis (TV) infection, Chlamydia trachomatis (CT) infection or gonococcal vaginitis;
2. History of systemic organic diseases or psychiatric diseases;
3. Planning for or during pregnancy, lactation, menstruation;
4. within 5 days of onset of the disease, any antibiotics has been used;
5. Long-term use of contraceptives or immunosuppressant;
6. Anaphylactic constitution or allergic to known ingredients of research drugs.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruifang Wu, M.D., Study Director — Dept of Obstetrics and Gynecology,Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women who came to the gynaecological clinic of Peking University Shenzhen Hospital, China, between March 2019 and June 2019 with abnormal vaginal discharge symptoms were recruited.
Period: Overall Study
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
Started | 63 | 63
Completed | 52 | 47
Not Completed | 11 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 2 | 1
Not completed — Protocol Violation | 3 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Complain of the research staff and refused to continue the trial | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal | Total
Number analyzed (Participants) | 52 | 47 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (7.0) | 33.3 (7.5) | 33.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 47 | 99
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 52 | 47 | 99
Employment status [Count of Participants; unit: Participants]
  Stable job | 43 | 41 | 84
  Unemployed or unstable work | 9 | 6 | 15
Smoking [Count of Participants; unit: Participants] | 5 | 2 | 7
Current relationship status [Count of Participants; unit: Participants]
  Married | 36 | 26 | 62
  Single, divorced or separated | 16 | 21 | 37
Childbirth history [Count of Participants; unit: Participants]
  At least one previous birth | 31 | 26 | 57
  No birth before | 21 | 21 | 42
Sexual activity [Count of Participants; unit: Participants]
  Sexual activity (vaginal sex) ≥ 3 times per one month | 28 | 20 | 48
  Had no sexual activity in the last half of the year or vaginal sex less than 3 times per one month | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Related Clinical Signs or Symptoms at Baseline
Description: Clinical signs and symptoms of bacteria vaginosis (BV), including homogeneous and thin vaginal discharge, unpleasant odour (such as a "fishy" smell) and vulvar discomfort (such as itching or burning), were recorded at baseline, the number of participants with related clinical signs or symptoms at Baseline were calculated.
Time Frame: 1 day before starting treatment
Population: Full analysis set of all randomized participants, that is 126, who had baseline samples were tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
Number analyzed (Participants) | 63 | 63
Participants | 63 | 63
Statistical Analysis 1: Comparison: Probiotics and Metronidazole vs Metronidazole Vaginal; Test type: Non-Inferiority — The relevant parameters were determined as follows: test level α=0.05, test power 1-β=0.80, Pt=0.90, Pc=0.75, Nt:Nc=1:1, boundary value Δ= -0.0.068 (excellent), and Fisher's exact test. As a result, the sample size of each group was calculated as 50 patients, 100 patients in total. Considering a loss to follow-up rate of 20%, a sample size of 120 patients was finally determined, with 60 patients in each group; p < 0.01, Chi-squared

2. Primary Outcome: Number of Participants With Clinically Effective in Each Study Arm in the 30-day Follow-up
Description: Clinical signs and symptoms of BV, including homogeneous and thin vaginal discharge, unpleasant odour (such as a "fishy" smell) and vulvar discomfort (such as itching or burning), were recorded at the 30-day, the number of participants with clinically effective (with the sign or symptoms disappeared or released compared with the baseline data) were calculated.
Time Frame: the 30th day after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
Number analyzed (Participants) | 52 | 47
Participants | 30 | 28
Statistical Analysis 1: Comparison: Probiotics and Metronidazole vs Metronidazole Vaginal; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.01, Chi-squared

3. Primary Outcome: Number of Participants With Clinically Effective in Each Study Arm at the 90-day Follow-up
Description: Clinical signs and symptoms of BV, including homogeneous and thin vaginal discharge, unpleasant odour (such as a "fishy" smell) and vulvar discomfort (such as itching or burning), were recorded at the 30-day, the number of participants with clinically effective (with the sign or symptoms disappeared or released compared with the 30-day follow-up data) were calculated.
Time Frame: the 90th day after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
Number analyzed (Participants) | 30 | 28
Participants | 19 | 23
Statistical Analysis 1: Comparison: Probiotics and Metronidazole vs Metronidazole Vaginal; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.01, Chi-squared

4. Primary Outcome: Number of Participants With Bacteriological Cure in Each Study Arm at the 30-day Follow-up
Description: A vaginal swab for bacteriological assessment of BV by Nugent criteria was performed. The Nugent score can range from 0 to 10. Bacteriological cure of BV was defined as a normal Nugent score of 0-6. Participants who were clinical failures, or had a Nugent score ≥ 7 were therapeutic failures.
Time Frame: the 30th day after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
Number analyzed (Participants) | 52 | 52
Participants | 30 | 28
Statistical Analysis 1: Comparison: Probiotics and Metronidazole vs Metronidazole Vaginal; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.01, Chi-squared

5. Primary Outcome: Number of Participants With Bacteriological Cure in Each Study Arm at the 90-day Follow-up
Description: as for outcome 4
Time Frame: the 90th day after starting treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
Number analyzed (Participants) | 30 | 28
Participants | 19 | 23
Statistical Analysis 1: Comparison: Probiotics and Metronidazole vs Metronidazole Vaginal; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality and Serious Adverse Events were monitored/assessed, but none were observed.
Arm/Group | Probiotics and Metronidazole | Metronidazole Vaginal
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 5/63 | 6/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Probiotics and Metronidazole (N=63) | Metronidazole Vaginal (N=63)
vaginal itching or burning (Infections and infestations) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03894813/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03894813/ICF_001.pdf